CLINICAL TRIAL: NCT06688864
Title: Delivery of an eHealth Intervention for Under-resourced Adults With Chronic Pain (Flourish Study)
Brief Title: Under-Resourced Adults With Chronic Pain eHealth Study
Acronym: Flourish
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Eleshia Morrison, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 23-009761
Record Dates: First submitted 2024-11-13; First posted 2024-11-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Black adults with chronic pain (Experimental)
  Interventions: Behavioral: EPIO App
- LGBTQIA+ adults with chronic pain (Experimental)
  Interventions: Behavioral: EPIO App

INTERVENTIONS:
Behavioral: EPIO App — Participants will receive access to the app-based cognitive-behavioral pain self-management intervention program (EPIO) for 3 months.

SUMMARY:
The purpose of this study is to examine the feasibility of the dissemination of a cognitive-behavioral eHealth application (app) for pain self-management with Black and LGBTQ+ adults with high-impact chronic pain lasting at least 3 months and disrupting daily functioning (Implementation aim).

ELIGIBILITY:
Inclusion Criteria:

* Identify as Black or LGBTQ+.
* Reside in MN, WI, or IA.
* Chronic pain diagnosis for at least 3 months.
* Experience chronic pain that makes it harder to do their day-to-day activities
* Have daily access to a smart mobile device (smartphone or table) and are willing to use the EPIO app.

Exclusion Criteria:

* Unable or unwilling to use the digital app for the study
* Do not have daily access to a smart mobile device (smartphone or tablet)
* Self-report cancer related pain, or severe untreated psychological illness (e.g., psychosis); and/or do not fit into one of the demographic categories listed in #1-3 for inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-07-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in West Haven Yale Multiphasic Pain Inventory (WHYMPI) score | Baseline, 3 months
  The West Haven Yale Multiphasic Pain Inventory (WHYMPI) is a 52-item measure of various domains of the experience of pain, including pain interference (primary intervention outcome) and pain severity with daily functioning.

SECONDARY OUTCOMES:
Change in Pain Catastrophizing Scale (PCS) score | Baseline, 3 months
  The Pain Catastrophizing Scale (PCS) is a self-report questionnaire designed to assess catastrophic thinking related to pain. It consists of 13 items, each rated on a 5-point scale from 0 (not at all) to 4 (all the time). The total score ranges from 0 to 52, with higher scores indicating greater levels of catastrophizing.
Change in Pain Self-Efficacy Questionnaire (PSEQ) score | Baseline, 3 months
  The Pain Self-Efficacy Questionnaire (PSEQ) is a 10-item questionnaire developed to assess the confidence people with ongoing pain have in performing activities while in pain. A raw score is presented with a range from 0 - 60, where high scores indicate greater levels of confidence in dealing with pain.
Change in Chronic Pain Acceptance Questionnaire-Revised (CPAQ-R) score | Baseline, 3 months
  The Chronic Pain Acceptance Questionnaire (CPAQ-R) consists of 20 items, with 10 items each for the subscales of Activity Engagement and Pain Willingness. The items on the CPAQ are rated on a 7-point scale from 0 (never true) to 6 (always true). Higher scores indicate higher levels of acceptance.
Change in Hospital Anxiety and Depression Scale (HADS) score | Baseline, 3 months
  The Hospital Anxiety and Depression Scale is a 14-item scale with seven items each for the anxiety and depression symptom subscales. For both subscales, a score of 8-10 indicates mild symptoms, 11-14 indicates moderate symptoms, and 15-21 indicates severe symptoms.
Change in Short Form-36 score | Baseline, 3 months
  The SF-36 Health Survey is a 36-item, participant-reported survey that measures patient health and disability. Possible scores range from 0 to 100, with 0 indicating maximum disability, and 100 indicating no disability.
Change in Alcohol Use Disorders Identification Test-Concise (AUDIT-C) score | Baseline, 3 months
  The AUDIT-C consists of three questions, and each question has 5 answer choices valued from 0 points to 4 points. The AUDIT-C is scored on a scale of 0-12. A score of 4 for men and a score of 3 for women can raise suspicion of alcohol use disorder.
Change in Perceived Stress Scale (PSS) score | Baseline, 3 months
  The 10-item Perceived Stress Scale (PSS) measures global perceived stress experienced by the participant over the preceding 30 days. The questions in this assessment tool ask how often the participant felt or thought a certain way during the past month. Possible answers include: 0 - never; 1 - almost never; 2 - sometimes; 3 - fairly often, and 4 - very often. Possible scores range from 0 to 40, with lower scores indicating a better outcome (less stress).
System Usability Scale score (SUS) | 3 months
  The System Usability Scale is a 10-item measure of overall usability of the app regarding perceived usefulness and ease of use. The overall score is in a range from 0-100, with a higher score indicating better user satisfaction.
Everyday Discrimination Scale-Expanded (EDS-E) score | Baseline
  The Everyday Discrimination Scale-Expanded (EDS-E) is a self-report measure used to assess the frequency of various forms of discrimination experienced by individuals in their day-to-day lives. It consists of 10 items, each rated on a 5-point Likert scale from 0 (never) to 4 (very often).

CONTACTS AND LOCATIONS:
Overall Officials: Eleshia J. Morrison, Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No